CLINICAL TRIAL: NCT03144349
Title: Is Variation of Plasmatic Protein Concentration During Continuous Renal Replacement Therapy Predictive of Hypovolemia in Intensive Care Unit?
Brief Title: Diagnosis Accuracy of Hemoconcentration to Detect Hypovolemia During CRRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hopital Louis Pradel (Other)
Responsible Party: Principal Investigator, Matthias Jacquet-Lagrèze, Medical Doctor, Hopital Louis Pradel
Other Study IDs: 2016-A01830-51
Record Dates: First submitted 2016-12-26; First posted 2017-05-08 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Continuous Renal Replacement Therapy; Intensive Care Unit; Hypovolemia; Fluid Overload
MeSH Terms: conditions — Hypovolemia; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Ionogram Protidemia Hemogram
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to analyze if blood protein concentration variation during continuous renal replacement therapy (CRRT) with fluid removal can predict a decrease of 15 % of cardiac index in intensive care unit (ICU) patients. Blood protein concentration, clinical data describing hemodynamic status (providing data from Pulsion medical system PiCCO2 ® monitoring), including preload dependency evaluation with passive leg raising, are collected at different times: before initiation of fluid removal, and after the first episode of hypotension or one hour after initiation of fluid removal.

DETAILED DESCRIPTION:
The aim of the study is to analyze if blood protein concentration variation during continuous renal replacement therapy (CRRT) with fluid removal can predict a decrease of 15 % of cardiac index in intensive care unit (ICU) patients. Blood protein concentration, clinical data describing hemodynamic status (providing data from Pulsion medical system PiCCO2 ® monitoring), including preload dependency evaluation with passive leg raising, are collected at different times: before initiation of fluid removal, and after the first episode of hypotension or one hour after initiation of fluid removal.

ELIGIBILITY:
Inclusion Criteria:

* up to 18 years old
* continuous renal replacement therapy
* Suspicion of fluid overload
* Prescription of fluid removal by the intensivist
* PICCO2 monitoring

Exclusion Criteria:

* pregnancy
* intra abdominal hypertension
* Moribund patient
* Abdominal hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have PiCCO2 ® monitoring and continuous renal replacement therapy with a prescription of fluid removal in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
plasmatic protein concentration variation | 1 hour
  Two sample of plasmatic protein before and after a fluid removal will be performed. The variation of the protein concentration (computed as the difference between final and baseline value divided by the baseline value expressed in %) will be the index test to diagnose a decrease of cardiac output of more than 15 % due to the fluid removal.

SECONDARY OUTCOMES:
Plasmatic protein concentration in patient with preload dependency before fluid removal | 1 hour
  hemoconcentration will be evaluated in the subgroup of preload dependent patients
Central venous pressure (CVP) | 1 hour
  CVP will be tested to evaluate the diagnostic ability to diagnose a reduction of cardiac output due the fluid removal
Global end diastolic volume (GEDV) | 1 hour
  GEDV, calculated with transpulmonary thermodilution will be tested to evaluate the diagnostic ability to diagnose a reduction of cardiac output due the fluid removal
Extravascular lung water (EVLW) | 1 hour
  EVLW, calculated with transpulmonary thermodilution will be tested to evaluate the diagnostic ability to diagnose a reduction of cardiac output due the fluid removal
hemoconcentration evaluated with hemoglobin variation | 1 hour
  hemoconcentration evaluated with hemoglobin variation will be tested to evaluate the diagnostic ability to diagnose a reduction of cardiac output due the fluid removal

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Fellahi, M.D.,Ph.D., Study Director — Hopital Louis Pradel
Locations (2):
- France (2):
  - Hôpital Cardiologique Louis Pradel, Lyon, Auvergne-Rhône-Alpes
  - Matthias Jacquet-Lagreze, Lyon, Rhône

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lamia B, Ochagavia A, Monnet X, Chemla D, Richard C, Teboul JL. Echocardiographic prediction of volume responsiveness in critically ill patients with spontaneously breathing activity. Intensive Care Med. 2007 Jul;33(7):1125-1132. doi: 10.1007/s00134-007-0646-7. Epub 2007 May 17. PMID 17508199
- [Background] Monnet X, Marik P, Teboul JL. Passive leg raising for predicting fluid responsiveness: a systematic review and meta-analysis. Intensive Care Med. 2016 Dec;42(12):1935-1947. doi: 10.1007/s00134-015-4134-1. Epub 2016 Jan 29. PMID 26825952
- [Background] Monnet X, Cipriani F, Camous L, Sentenac P, Dres M, Krastinova E, Anguel N, Richard C, Teboul JL. The passive leg raising test to guide fluid removal in critically ill patients. Ann Intensive Care. 2016 Dec;6(1):46. doi: 10.1186/s13613-016-0149-1. Epub 2016 May 20. PMID 27207178
- [Background] Bitker L, Bayle F, Yonis H, Gobert F, Leray V, Taponnier R, Debord S, Stoian-Cividjian A, Guerin C, Richard JC. Prevalence and risk factors of hypotension associated with preload-dependence during intermittent hemodialysis in critically ill patients. Crit Care. 2016 Feb 23;20:44. doi: 10.1186/s13054-016-1227-3. PMID 26907782